CLINICAL TRIAL: NCT00902889
Title: Single Centre (Pilot) Study for Deep Brain Stimulation (DBS) of the Globus Pallidus in Huntington's Disease (HD)
Brief Title: Deep Brain Stimulation of the Globus Pallidus in Huntington's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Huntington
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Huntington's Disease
Keywords: Globus pallidus; Huntington's Disease; Deep Brain Stimulation; Movement Disorders
MeSH Terms: conditions — Huntington Disease; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 6 weeks stimulation with GPI (lower caudal two contacts), 4 weeks wash-out, 6 weeks stimulation with GPE (upper cranial two contacts).
  Interventions: Procedure: Stimulation
- 2 (Experimental): 6 weeks stimulation with GPE (upper cranial two contacts), 4 weeks wash-out, 6 weeks stimulation with GPI (lower caudal two contacts)
  Interventions: Procedure: Stimulation

INTERVENTIONS:
Procedure: Stimulation — 6 weeks stimulation with GPI (lower caudal two contacts), 4 weeks wash-out, 6 weeks stimulation GPE (upper cranial two contacts)
  Other Names: GPI; GPE
  Arms: 1
Procedure: Stimulation — 6 weeks stimulation with GPE (upper cranial two contacts), 4 weeks wash-out, 6 weeks stimulation with GPI (lower caudal two contacts)
  Other Names: GPE; GPI
  Arms: 2

SUMMARY:
This is a single centre, controlled phase I study, which evaluates safety and efficacy of stimulation of lower caudal two contacts (GPI) vs. upper cranial two contacts (GPE) in Huntington´s disease (HD).

DETAILED DESCRIPTION:
A total of 6 HD patients will be selected out of an existing larger HD patient cohort upon careful evaluation of the inclusion and exclusion criteria at month 0. Patients will be recruited if no significant cognitive deterioration is observed between month 0 and month 3. The preoperative clinical status will be evaluated twice including the United Huntington Disease Rating Scale (UHDRS), neuropsychological, neurophysiologic and neuroradiological assessments. At 4 weeks postoperatively an extensive evaluation of effects and side effects of every single contact of the bilateral quadripolar electrodes takes place.

All patients will receive a stereotactic placement of bilateral stereotactic insertion of two quadripolar electrodes into the Globus pallidus, two contacts reaching the GPE, two the GPI within both hemispheres. Surgery will be done under general anesthesia, The implantation of the stimulator (Kintera®) will take place in the same procedure. Postoperatively patients will be monitored at three and six months and regularly up to 60 months with a battery of clinical, neuropsychological, psychiatric, neurophysiological and neuroimaging tests.

We expect that this trial will provide a rational basis to conclude about the efficacy, safety, reproducibility and long-term effects of pallidal Deep Brain Stimulation (DBS) on motor symptoms of HD.

ELIGIBILITY:
Inclusion Criteria:

* clinically symptomatic and genetically confirmed Huntington Disease (number of CAG repeats>= 36)
* age: > 18
* moderate stage of the disease (UHDRS motor>= 30)
* predominant movement disorder
* compliance of the patient, stable cognition during a 6 months phase prior to inclusion (MDS>/= 120)
* signed informed consent

Exclusion Criteria:

* advanced disease, precluding the ability to give informed consent
* very early stage of disease causing minor disability
* severe comorbidity that could compromise the life prognostic or preclude general anaesthesia or immunosuppression
* Mattis Dementia Rating Scale < 120
* psychiatric or personality disturbances that might compromise the follow-up
* participation at another trial (in particular transplantation)
* severe cortical atrophy seen on CT and MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of stimulation of GPI versus GPR (UHDRS Scale) | 3 months after stimulation treatment

SECONDARY OUTCOMES:
Effect of treatment on cognitive functions (neuropsychological tests) | 3 months after stimulation treatment
Effects of treatment on electrophysiological tests | 3 months after stimulation treatment
Effects of treatment on functional scale (functional ability, dependence scale, TFC) | 3 months after stimulation treatment
Progression of disease (motor UHDRS) | 12 months after stimulation treatment
Effect of treatment on striatal atrophy (CT Scans) | 3 months after stimulation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vesper, Prof. Dr., Principal Investigator — Functional Neurosurgery and Stereotaxy, Department of Neurosurgery
Locations (1):
- Functional Neurosurgery and Stereotaxy, Department of Neurosurgery University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Temel Y, Cao C, Vlamings R, Blokland A, Ozen H, Steinbusch HW, Michelsen KA, von Horsten S, Schmitz C, Visser-Vandewalle V. Motor and cognitive improvement by deep brain stimulation in a transgenic rat model of Huntington's disease. Neurosci Lett. 2006 Oct 2;406(1-2):138-41. doi: 10.1016/j.neulet.2006.07.036. Epub 2006 Aug 14. PMID 16905252
- [Derived] Ferrea S, Groiss SJ, Elben S, Hartmann CJ, Dunnett SB, Rosser A, Saft C, Schnitzler A, Vesper J, Wojtecki L; Surgical Approaches Working Group of the European Huntington's Disease Network (EHDN). Pallidal deep brain stimulation in juvenile Huntington's disease: local field potential oscillations and clinical data. J Neurol. 2018 Jul;265(7):1573-1579. doi: 10.1007/s00415-018-8880-1. Epub 2018 May 3. PMID 29725840
- [Derived] Beste C, Muckschel M, Elben S, J Hartmann C, McIntyre CC, Saft C, Vesper J, Schnitzler A, Wojtecki L. Behavioral and neurophysiological evidence for the enhancement of cognitive control under dorsal pallidal deep brain stimulation in Huntington's disease. Brain Struct Funct. 2015 Jul;220(4):2441-8. doi: 10.1007/s00429-014-0805-x. Epub 2014 May 31. PMID 24878825